CLINICAL TRIAL: NCT00928902
Title: Pilot Phase II Trial for the Evaluation of the Effect of Systemic Low-dose IL-2 on the Immunogenicity of a Vaccine Comprising Synthetic Melanoma Peptides Administered With GM-CSF-in-Adjuvant, in Patients With High Risk Melanoma
Brief Title: Trial for the Evaluation of the Effect of Systemic Low-dose Interleukin-2 (IL-2) on the Immunogenicity of a Vaccine Comprising Synthetic Melanoma Peptides Administered With Granulocyte-macrophage Colony-stimulating Factor (GM-CSF)-In-Adjuvant, in Patients With High Risk Melanoma
Acronym: MEL36
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Craig L Slingluff MD, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 8515
Record Dates: First submitted 2009-06-24; First posted 2009-06-26 (Estimated); Last update posted 2010-10-21 (Estimated); Status verified 2010-10

CONDITIONS: Melanoma
Keywords: melanoma; vaccine; peptides; adjuvant; immunogenicity; stage IIB, stage III or resected stage IV
MeSH Terms: conditions — Melanoma | interventions — Interleukin-2; polyvalent melanoma cell vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Peptides with GM-CSF-in-adjuvant, with upfront IL-2 (Active Comparator): Each of the peptides plus tetanus toxoid peptide, plus GM-CSF in adjuvant, administered subcutaneously and intradermally. Systemic low-dose IL-2 will be administered daily for 6 weeks, beginning at week 1 and ending at week 7.
  Interventions: Drug: low-dose IL-2; Biological: melanoma vaccine
- Peptides plus GM-CSF-in-adjuvant, delayed IL-2 (Active Comparator): Peptides plus GMCSF-in-adjuvant, with delayed IL-2.
  Each of the peptides plus tetanus toxoid peptide, plus GM-CSF in adjuvant, administered subcutaneously and intradermally. Systemic low-dose IL-2 will be administered daily for 6 weeks, beginning at week 4 and ending at week 10.
  Interventions: Drug: low-dose IL-2; Biological: melanoma vaccine

INTERVENTIONS:
Drug: low-dose IL-2 — low-dose IL-2, administered daily for 6 weeks, to begin either at week 1 (group 1) or week 4 (group 2)
Biological: melanoma vaccine — six melanoma vaccines given over a 6-week period

SUMMARY:
This clinical pilot study will test the hypothesis that systemic low-dose IL-2 therapy significantly enhances the immunologic efficacy of a vaccine comprising melanoma peptides plus GM-CSF-in-adjuvant.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have been diagnosed, by cytologic or histologic examination, with AJCC stage IIB, stage III or resected stage IV melanoma.
* Patients with up to 2 brain metastases less than or equal to 2 cm that have been surgically removed or treated successfully with the gamma-knife are eligible. Surgical resections must have been performed within 6 months prior to entry.
* All patients must have:

  1. ECOG performance status 0-1, and,
  2. Ability and willingness to give informed consent.
* Laboratory parameters as follows:

  * HLA-A1, A2 or A3 (+)
  * gp100 (+) and/or tyrosinase (+) tumor cells
  * ANC > 1000/mm3, and Platelets > 100,000 and Hgb > 9
  * Hepatic: AST and ALT up to 2.5 x upper limits of normal (ULN), Bilirubin up to 2.5 x ULN, Alkaline phosphatase up to 2.5 x ULN
  * Renal: Creatinine up to 1.5 x ULN
  * Serology: HIV negative, Hepatitis C negative

Exclusion criteria:

* Patients who are currently receiving cytotoxic Chemotherapy or radiation or who have received that therapy within the preceding 4 weeks.
* Patients with known or suspected allergies to any component of the vaccine.
* Patients receiving the following medications at study entry or within the preceding 30 days are excluded:

  * Agents with putative immunomodulating activity (with the exception of non-steroidal anti-inflammatory agents)
  * Allergy desensitization injections
  * Corticosteroids, administered parenterally or orally - topical corticosteroids are acceptable
* Any growth factors, Interleukin 2, Interferon alfa.
* Prior melanoma vaccinations will not be an exclusion criteria if given more than 8 weeks previously, but will be recorded, and data analysis will take this into account.
* Other investigational drugs or investigational therapy also will not necessarily be an exclusion criteria, but will similarly be recorded and taken into account during data analysis.
* Pregnancy or the possibility of becoming pregnant during vaccine administration.

  * Female patients of child-bearing potential must have a negative pregnancy test (urinary or serum beta-HCG) prior to administration of the first vaccine dose.
  * Males and females must agree, in the consent form, to use effective birth control methods during the course of vaccination.
  * This is consistent with existing standards of practice for vaccine and chemotherapy protocols.
* Patients in whom there is a medical contraindication or potential problem in complying with the requirements of the protocol, in the opinion of the investigator.
* Patients classified according to the New York Heart Association classification system as having Class II, III or IV heart disease.
* Patients with active connective tissue disease requiring medication, or other severe autoimmune disease.
* Patients who are actively hyperthyroid.
* Patients with uncontrolled diabetes.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 1999-11; Primary Completion 2001-04 (Actual); Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
To evaluate the effect of systemic low-dose IL-2 on the immunogenicity of a vaccine comprising synthetic melanoma peptides plus GM-CSF-in-adjuvant.

SECONDARY OUTCOMES:
Changes in disease, analysis of melanoma antigen (gp100, tyrosinase, MART-1) expression on melanoma cells from metastatic sites, Vitiligo.

CONTACTS AND LOCATIONS:
Overall Officials: Craig L Slingluff, MD, Principal Investigator — University of Virginia